CLINICAL TRIAL: NCT01908491
Title: Comparison of the Effects of Opioid-Based Intravenous Patient Controlled Analgesia and Continuous Ropivacaine Infusion Through Wound Catheters After Repair of Pectus Excavatum
Brief Title: Comparison of IV PCA and Wound Infusion After Repair of Pectus Excavatum
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: The Catholic University of Korea (Other)
Responsible Party: Principal Investigator, Jeong Eun Kim, Clinical Assistant Professor, The Catholic University of Korea
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: pectus-pain study
Record Dates: First submitted 2013-07-19; First posted 2013-07-25 (Estimated); Last update posted 2013-11-14 (Estimated); Status verified 2013-11

CONDITIONS: Pain; Side Effects
Keywords: patient controlled analgesia; wound catheter infusion; postoperative pain control; pectus excavatum; pain score
MeSH Terms: conditions — Pain; Funnel Chest | interventions — Analgesia, Patient-Controlled

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- IV PCA (Active Comparator): hydromorphone with ketorolac
  Interventions: Device: IV PCA
- Continuous wound infusion (Experimental): ON-Q Painbuster with ropivacaine
  Interventions: Device: Continuous wound infusion

INTERVENTIONS:
Device: IV PCA — On arrival in the postanesthetic care unit, a patient-controlled analgesia (IV PCA) was connected to the iv catheter. The PCA regimen consisted of hydromorphone (2 mcg/kg/hr) and ketorolac (0.02 mg/kg/hr) with normal saline (total volume 100ml). PCA was programmed to deliver 1 ml/hr as background infusion and 1 ml per demand with a 10 min lockout during 48 hr period.
  Arms: IV PCA
Device: Continuous wound infusion — Patients underwent insertion of wound catheters by the surgeon just before the closure of incision site. The wound catheters, consisting of double branch and connected to elastomeric pump filled with ropivacaine (0.15~0.25%) and administered at a constant flow rate of 2 ml/hr in each branch of the catheter for 48 hr.
  Arms: Continuous wound infusion

SUMMARY:
Postoperative pain management is a major problem after repair of pectus excavatum.Various methods of pain management have been introduced. However, the effects of continuous wound infusion of local anesthetics through ON-Q catheters were not well evaluated in pectus surgery. Therefore, we conducted prospective randomized controlled study to compare the effects of IV PCA and continuous wound infusion after repair of pectus excavatum.

DETAILED DESCRIPTION:
Pain control is an important issue after correction of pectus excavatum. Insufficient pain control leads to develop postoperative pulmonary complications, such as hypoxia, atelectasis and pneumonia. Additionally, hospital length of stay could be prolonged. Therefore, successful pain management is mandatory to improve clinical outcome, to decrease postoperative morbidity and to shorten the duration of hospital stay. Various methods of pain management have been introduced. Current typical methods for pain management include thoracic epidural analgesia and intravenous patient-controlled analgesia (IV PCA). Epidural analgesia has shown superior pain control effects. However, there may be rare but serious complications, such as spinal cord and nerve root lesions, epidural hematoma, or infections. IV PCA is a well-established method of postoperative pain management. However, the systemic side effects of opioid, such as nausea, vomiting, sedation, or respiratory depression may occur. Continuous wound infusion of local anesthetics through ON-Q catheters is another method for pain management. It has been used for various surgical procedures. However, the effect is not well evaluated in pectus surgery. The purpose of this study is to compare the effects of opioid-based IV PCA and continuous wound infusion using a catheter.

ELIGIBILITY:
Inclusion Criteria:

* patients undergoing the repair of pectus excavatum

Exclusion Criteria:

* allergy to opioid or local anesthetics
* reoperation

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2012-10; Primary Completion 2013-10 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
Changes of pain score | during 48 hours after surgery
  Pain score was measured by the Wong-Baker FACES pain scale at 1, 2, 6, 24, 48 hours after surgery. Pain scale consists of 6 faces with word descriptors and numbers from 0 to 10. The child look at the faces, the nurse or parent uses the words to describe the expression, and the child is asked to point to the face that describes how he/she feels. The number is used to record a pain score. This simple and quick scale can be easily reproduced for use at the bed-side with children as young as 3 years of age.

SECONDARY OUTCOMES:
Incidence of side effects | during 48 hours after surgery
  Number of patients who developed nausea, vomiting, sedation, respiratory depression,or wound catheter related complications are recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Jeong Eun Kim, MD, PhD, Principal Investigator — Seoul St. Mary's Hospital, the Catholic University of Korea
Locations (1):
- Seoul St. Mary's Hospital, the Catholic University of Korea, Seoul, South Korea